CLINICAL TRIAL: NCT05358405
Title: Prediction Of Pulmonary Edema With Müller Maneuver
Acronym: PoEM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study received an unfavorable opinion from the Ethics Committee to extend the study.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-A02864-53
Record Dates: First submitted 2022-03-14; First posted 2022-05-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Weaning; Spontaneous Breathing Trial
Keywords: Weaning; Spontaneous breathing trial; Pulmonary edema; Passive leg raising; Cardiac output; Müller maneuver
MeSH Terms: conditions — Pulmonary Edema

STUDY DESIGN:
Intervention Model Description: Diagnostic of weaning failure due to pulmonary edema
Masking Description: Experimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Müller maneuver (Other): Open Label with intervention Müller maneuver
  Interventions: Other: Müller maneuver

INTERVENTIONS:
Other: Müller maneuver — The Müller maneuver allows maximum inspiratory pressure measurement via a one-way valve connected to the intubation tube and is currently used in routine care for diaphragmatic assessment. Ventilation through the one-way valve results in forced inspiration for about 20 seconds. The endothoracic depression induced by this test is likely increasing venous return and cardiac output in patients with preload reserve, i.e. in preload-dependent patients. The observation of an increase in cardiac output during a Müller maneuver could reflect the existence of a dependent preload state, i.e. with a reserve of preload, and de facto lower risk of pulmonary oedema. This test would be an easy alternative to the passive leg raising test used in current practice to evaluate the preload dependency and the risk of weaning induced pulmonary edema.

SUMMARY:
The mechanical ventilation weaning must begin as early as possible to limit its complications and requires a spontaneous breathing trial (SBT) before the separation from the ventilator to the patient.

However, some patients fail this test and cannot be extubated. The main causes are pulmonary edema and diaphragmatic dysfunction. Predicting the risk of failure before carrying out the SBT makes it possible to anticipate a failure of the extubation and to adapt the therapies as well as possible. To assess the risk of pulmonary edema, cardiac preload, which corresponds to the end-diastolic filling volume of the ventricle, can be estimated using simple tests as the passive leg raising test before an SBT.

However, this test requires tilting the patient's trunk and raising the lower limbs to 45°, and is not practical, especially in intensive care.

The Müller maneuver, which allows maximum inspiratory pressure measurement via a one-way valve connected to the intubation tube, is currently used in routine care for diaphragmatic assessment. The endothoracic depression induced by this test is likely increasing venous return and cardiac output in patients with a reserve of preload, i.e. in preload-dependent patients. This test would be an easy alternative to the passive leg raising test used in current practice.

The objectif is to assess whether the presence of an independant prelaod state, as detected by the absence of increased cardiac output during the Müller maneuver, is associated with the occurence of pulmonary edema during weaning from mechanical ventilation.

The study consist in the measurement of cardiac output before and after the passive leg raising test and the Müller maneuver, then measurement of cardiac output before and after an SBT.

A transthoracic ultrasound and a blood sample with dosage of proteins and hemoglobin will be carried out initially and then at the end of the SBT as part of routine care.

The investigators hypothesize:

* The Müller maneuver induces a greater increase in cardiac output in patients in a state of preload dependancy than in patients in a state of preload independancy.
* The absence of documented preload dependancy during a Müller maneuver is associated with the occurrence of pulmonary edema during an SBT.

The investigators included patients :

* > 18 years old, conscious patient, with health insurance, placed under mechanical ventilation for at least 24 hours ;
* In whom it was decided to perform a passive leg raising test and an SBT. The investigators excluded pregnancy, patient with chest tube, particpation in another interventional study, tracheostomy, patient under legal protection.

DETAILED DESCRIPTION:
The mechanical ventilation weaning must begin as early as possible to limit its complications and requires a spontaneous breathing trial (SBT) before the separation from the ventilator to the patient. The main causes of weaning failure are pulmonary edema and diaphragmatic dysfunction. Predicting the risk of failure before carrying out the SBT makes it possible to anticipate a failure of the extubation and to adapt the therapies as well as possible.

To predict the risk of pulmonary edema, physician could 1/ estimate the cardiac preload, which corresponds to the end-diastolic filling volume of the ventricle, using simple tests as the passive leg raising test before an SBT. This test requires tilting the patient's trunk and raising the lower limbs to 45°, and is not practical, especially in intensive care 2/ measure the hemoconcentration (hemoglobin and protein variation before and after SBT). However, this tests are not easy in intensive care unit.

The Müller maneuver, which allows maximum inspiratory pressure measurement via a one-way valve connected to the intubation tube, is currently used in routine care for diaphragmatic assessment. The endothoracic depression induced by this test is likely increasing venous return and cardiac output in patients with a reserve of preload, i.e. in preload-dependent patients. This test would be an easy alternative to the passive leg raising test used in current practice.

The objectif is to assess whether the presence of an independant prelaod state, as detected by the absence of increased cardiac output during the Müller maneuver, is associated with the occurence of pulmonary edema during weaning from mechanical ventilation. The investigators include patients:

* Placed under mechanical ventilation for at least 24 hours ;
* In whom it was decided to perform a leg lift test and an SBT. Patients are intubated and ventilated on the ventilators of the intensive care unit (v500, Dräger Medical, Lübeck, Germany or Carescape r860, GE Healthcare, Buc, France). The initial settings are decided by the physician in charge of the patient according to the gas exchanges.

The passive leg raising test consists of transferring a patient from a semi-sitting position to a position in which the trunk is horizontal and the lower limbs are elevated at 45°. This is achieved by the electrically operated bed. The test is considered positive (preload dependency) if the cardiac output increases more than 10%. This test is performed in common practice to assess the cardiac preload of patients before an SBT. The cardiac output is measured by transpulmonary thermodilution (if the patient is equiped by this dispositif before the study) or by cardiac echography.

SBT consists of reproducing the ventilation conditions once the patient has been extubated. This test is carried out using a so-called "T" piece connected to the end of the intubation tube or by canceling the assistance of the ventilator during 30 minutes. This test is performed daily in intensive care in the intubated patient before any extubation.The determination of hemoglobin and plasma proteins consists of a blood sample via a catheter already in place and its analysis before and after the SBT. An increase in hemoglobin or plasmatique proteins by 6% detect a weaning pulmonary edema .

The acts/procedures added by the search are:

* Transthoracic ultrasound added for research if the monitoring system PiCCO2 is not set up in the patient as part of the treatment. Transthoracic echocardiography is a medical imaging technique based on the use of ultrasound, inaudible, painless and harmless sound waves that allow visualization of the cardiac silhouette, its functioning and allows measurement of cardiac output, fraction ventricular ejection and other diagnostic parameters for left heart failure and pulmonary edema (E/A and E/e' ratios). This technique is used in routine daily practice by physicians in charge of patient.
* Performing a Müller maneuver after the passive leg raising test. The Müller maneuver is used in current practice for measuring the maximum inspiratory pressue before performing an SBT. It consists of using a one-way valve connected to the intubation tube allowing forced inspiration with a closed glottis, and lasts about twenty seconds.
* Measurement of cardiac output before and after a passive leg raisong, a Müller maneuver and an SBT.

Since the observation of cardiac output during the Müller maneuver is not taken into account for the management of patients suitable for research, the research will not be able to lead to a direct benefit for the participants.

On the other hand, in the event of positive results of the study, a collective benefit is expected.

ELIGIBILITY:
Inclusion Criteria :

* Men and women over 18 years old ;
* With health insurance ;
* Placed under mechanical ventilation for at least 24 hours ;
* Conscious patient.

Exclusion Criteria:

* Pregnancy (blood assay of βHCG) ;
* Participation in another intervention study ;
* Patient with chest tube
* Tracheostomy ;
* Patient under legal protection ;
* Patient receiving state medical assistance (AME).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-09 (Estimated); Primary Completion 2024-05-09 (Estimated); Study Completion 2024-07-09 (Estimated)

PRIMARY OUTCOMES:
Number of pulmonary edema during an spontaneous breathing trial (SBT) | During the spontaneous breathing trial (SBT)
  Occurrence of pulmonary edema during an SBT as defined by :
  * A failure of the SBT defined by objective and subjective signs defined by Boles et al (signs of respiratory distress, agitation, cyanosis, tachycardia > 140 beats per minute, hypertension Pas > 180mmHg, respiratory rate > 35 cycles per minute) AND
  * One or both of the following criteria :
    * Ultrasound markers: E/e' ratio ≥ 13 + E/A ≥ 2
    * Hemoconcentration markers (≥ 6% increase in plasma proteins or hemoglobin) The E/A and E/e' ratios are calculated automatically by the ultrasound machine.
  The increase in proteins, and plasma hemoglobin are calculated according to the following formula:
  Increase in plasma proteins and hemoglobin, (%) = ((final value - initial value) / initial value) x 100

SECONDARY OUTCOMES:
Cardiac index before and after a passive leg raising test and a Müller maneuver | 1 minute before and during a passive leg raising test (when it induces its maximum effect, usually within a minute) and a Müller maneuver (when it induces its maximum effects, usually within 20 seconds)
  A positive spontaneous breathing trial (SBT) is defined by an increase of cardiac output > 10% ((value after-value before/value before))x100.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra BEURTON, MD, Principal Investigator — Pitié-Salpêtrière Hospital
Locations (1):
- Pitié-Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No